CLINICAL TRIAL: NCT00098982
Title: Phase I Study of PS-341 (VELCADE) in Combination With 5FU/LV Plus Oxaliplatin in Patients With Advanced Colorectal Cancer
Brief Title: Bortezomib, Fluorouracil, Leucovorin, and Oxaliplatin in Treating Patients With Advanced or Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: EORTC-16029; EORTC-16029; MILLENNIUM-EORTC-16029; 2004-001763-21 (EudraCT Number)
Record Dates: First submitted 2004-12-08; First posted 2004-12-09 (Estimated); Last update posted 2013-06-12 (Estimated); Status verified 2013-06

CONDITIONS: Colorectal Cancer
Keywords: stage III colon cancer; stage IV colon cancer; stage III rectal cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Bortezomib; Fluorouracil; Leucovorin; Oxaliplatin

INTERVENTIONS:
Drug: bortezomib
Drug: fluorouracil
Drug: leucovorin calcium
Drug: oxaliplatin

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as fluorouracil, leucovorin, and oxaliplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Bortezomib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. It may also help the chemotherapy drugs work better by making tumor cells more sensitive to the drugs. Giving bortezomib with fluorouracil, leucovorin, and oxaliplatin may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of bortezomib when given with fluorouracil, leucovorin, and oxaliplatin in treating patients with advanced or metastatic colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the dose-limiting toxicity and maximum tolerated dose of bortezomib when administered with fluorouracil, leucovorin calcium, and oxaliplatin in patients with advanced or metastatic colorectal cancer.
* Determine the recommended phase II dose of bortezomib in patients treated with this regimen.

Secondary

* Determine response in patients with measurable disease treated with this regimen.

OUTLINE: This is an open-label, non-randomized, multicenter, dose-escalation study of bortezomib.

Patients receive bortezomib IV over 3-5 seconds on days 1, 8, and 15; oxaliplatin IV over 2 hours on days 1 and 15; and leucovorin calcium IV over 2 hours and fluorouracil IV over 22 hours on days 1, 2, 15, and 16. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of bortezomib until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Additional patients receive treatment at the MTD to a maximum of 12 patients at that dose level.

Patients are followed every 8 weeks until disease progression or start of a new anticancer treatment.

PROJECTED ACCRUAL: Not specified.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed advanced or metastatic colorectal cancer
* Amenable to first-line treatment with oxaliplatin, fluorouracil, and leucovorin calcium for advanced or metastatic disease
* No symptomatic or radiologic evidence of brain metastases

PATIENT CHARACTERISTICS:

Age

* Over 18

Performance status

* ECOG 0-1

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count ≥ 2,000/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic

* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* Alkaline phosphatase ≤ 2.5 times ULN (5 times ULN if liver metastases are present)
* AST and ALT ≤ 2.5 times ULN (5 times ULN if liver metastases are present)

Renal

* Creatinine ≤ 1.7 mg/dL

Cardiovascular

* No ischemic heart disease within the past 6 months
* No clinically significant ECG changes

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No baseline neuropathy > grade 1
* No other prior or concurrent malignancy except cone-biopsied carcinoma of the cervix or adequately treated basal cell or squamous cell skin cancer
* No unstable systemic disease
* No active uncontrolled infection
* No psychological, familial, sociological, or geographical condition that would preclude study participation
* No hypersensitivity to bortezomib, boron, or mannitol

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior oxaliplatin
* No prior chemotherapy for advanced or metastatic disease
* At least 6 months since prior adjuvant chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* More than 4 weeks since prior radiotherapy

Surgery

* More than 14 days since prior major surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2004-09; Primary Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose and recommended dose of bortezomib as measured by CTC v3.0

SECONDARY OUTCOMES:
Safety as measured by CTC v3.0
Response as measured by RECIST every 8 weeks
Time to progression as measured by Kaplan Meier and RECIST every 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Caponigro, MD, Study Chair — Istituto Nazionale per lo Studio e la Cura dei Tumori
Locations (3):
- Istituto Nazionale per lo Studio e la Cura dei Tumori, Naples, Italy
- Centre Hospitalier Universitaire Vaudois, Lausanne, Switzerland
- Leeds Cancer Centre at St. James's University Hospital, Leeds, England, United Kingdom

REFERENCES:
- [Result] Caponigro F, Lacombe D, Twelves C, Bauer J, Govaerts AS, Marreaud S, Milano A, Anthoney A. An EORTC phase I study of Bortezomib in combination with oxaliplatin, leucovorin and 5-fluorouracil in patients with advanced colorectal cancer. Eur J Cancer. 2009 Jan;45(1):48-55. doi: 10.1016/j.ejca.2008.08.011. Epub 2008 Sep 20. PMID 18809314
- [Result] Lacombe DA, Caponigro F, Anthoney A, et al.: A phase I study of bortezomib in combination with 5FU/LV plus oxaliplatin in patients (pts) with advanced colorectal cancer (CRC): EORTC 16029. [Abstract] J Clin Oncol 25 (Suppl 18): A-4090, 2007.